CLINICAL TRIAL: NCT05399914
Title: Feasibility and Reliability of Synchronized Non-invasive Intermittent Positive Pressure Ventilation in Preterm Infants After Birth
Acronym: SenSyNoPP
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 310/2021BO1
Record Dates: First submitted 2022-04-20; First posted 2022-06-01 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2022-04

CONDITIONS: Preterm Infant; Delivery Room; Respiratory Support; Synchronized Noninvasive Positive Pressure Ventilation (SNIPPV)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Preterm infants with a gestational age (GA) between 26 ≥ and < 32 weeks
  Interventions: Other: S-NIPPV

INTERVENTIONS:
Other: S-NIPPV — Synchronized noninvasive positive pressure ventilation during the first 10 minutes after birth.

SUMMARY:
The aim of this prospective observational study (pilot study) is to test if synchronized noninvasive positive pressure ventilation (S-NIPPV) is feasible and works appropriately during transition from intrauterine to extrauterine life in very preterm infants in the delivery room.

DETAILED DESCRIPTION:
The study period will be the first 10 minutes after birth.

All patients will be non-invasively ventilated using an EVE NEO ventilator (CE 0482, Fritz Stephan GmbH, Gackenbach, Germany). A facemask will be used throughout the study period. Synchronization will be achieved using graseby capsule (Stephan, Vio Healthcare), which will be secured at the abdominal wall on the midaxillary line below the ribs. For the detection of spontaneous breaths respiratory induction plethysmography (RIP) is used. For this purpose, an extra small plethysmography belt (Sleepsense, Elgin, USA) is placed around the abdomen. The data of the plethysmography belts are processed and stored with the NewLifebox-XL (Advanced Life Diagnostics UG, Weener, Germany) and merged with the data from the ventilator for later evaluation.

Infants according to the clinician's assessment only needing CPAP will receive S-NIPPV with very low PIP levels. This enables to have enough ventilator breaths applied for analysis to obtain sufficient data about the synchronization rate of S-NIPPV in the delivery room and meanwhile consider the infant's safety by not applying high pressures where it might not be needed. The ventilator support settings will be PIP 10, PEEP 6 in the noninvasive pressure controlled assist control ventilation (nPC-ACV+) mode. In this mode every spontaneous breath is supported by a ventilator breath (if the triggering level is exceeded). The triggering level will be set at 0,5 to avoid autotriggering and unsupported breaths. The inspiratory time will be set at max. 0,3 sec. The backup ventilation rate is set at 60 per minute.The EVE NEO ventilator has in the nPC-ACV+ mode an option where the ventilator breaths are interrupted/stopped as soon as the graseby capsule detects a start of spontaneous expiration.

If the infant according to the clinician's assessment needs S-NIPPV (e.g. the infant is apnoeic, and/or heart rate is below 100 bpm), the pressure of S-NIPPV will be augmented to target PIP 20, PEEP 6 (unless clinical concerns require an adjustment). The respiratory support can be deescalated to PIP 10 once the clinician deems the higher pressure no longer necessary.

The following demographical characteristics will be collected from the patient charts (pseudonymized): gender, gestational age, birth weight, antenatal steroids, mode of delivery, reason for prematurity (prolong premature rupture of membrane, infection, pathologic CTG, pathological doppler, gestosis), time of cord clamping, umbilical cord pH, FiO2 requirement, APGAR.

The following interventions within the first 10 minutes after birth including the time will be noted: tactile stimulation, placement of an intravenous line, non-invasive surfactant administration, intubation, chest compression, administration of volume, catecholamine, blood or other medication.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a gestational age (GA) between 26 ≥ and < 32 weeks

Exclusion Criteria:

* Major congenital malformations
* Refused parental consent (prenatal parental consent is necessary)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants born at University Hospital in Tübingen.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Synchronisation rate | First 10 minutes after birth
  Synchronisation rate (sensitivity/true positive rate) of S-NIPPV in the delivery room meaning the proportion of graseby triggered synchronized ventilator breaths with corresponding RIP signal related to all spontaneous breaths detected by RIP.

SECONDARY OUTCOMES:
False negative rate | First 10 minutes after birth
  Proportion of non-synchronized ventilator breaths with corresponding RIP signal. This will be related to all spontaneous breaths detected by RIP.
False positive rate | First 10 minutes after birth
  Proportion of graseby triggered ventilator breaths without corresponding RIP signal. This will be related to all ventilator breaths without a corresponding RIP signal (i.e. movement artefacts).
Proportion of artifacts | First 10 minutes after birth
  Proportion of graseby triggered ventilator breaths without corresponding RIP signal. This will be related to all ventilator breaths.
Specificity (true negative rate) | First 10 minutes after birth
  Proportion of ventilator breaths without corresponding RIP signal and with no graseby signal (i.e. during an apnoea). This will be related to all ventilator breaths without a corresponding RIP signal.
Proportion of back up breaths | First 10 minutes after birth
  Proportion of ventilator breaths without corresponding RIP signal and with no graseby signal. This will be related to all ventilator breaths.
Proportion of time of synchronised breaths, non-synchronized breaths, periods of apnoea and periods of movement artefacts occure within the first ten minutes of respiratory support. | First 10 minutes after birth
Time until the graseby capsule is attached to the infant's abdomen and the proportion of infants in whom the graseby capsule is attached within the first two minutes after birth. | First 10 minutes after birth
Proportion of time non invasive ventilator breaths will be applied. | First 10 minutes after birth
Peak inspiratory pressure (PIP) | First 10 minutes after birth
Positive end expiatory pressure (PEEP) | First 10 minutes after birth
Mean airway pressure (MAP) | First 10 minutes after birth
Td (time delay) graseby | First 10 minutes after birth
  Time between the initial increase of the abdominal RIP curve and the initial increase of the graseby curve.
Td (time delay) ventilator | First 10 minutes after birth
  Time between the initial increase of the graseby curve and the beginning of the pressure curve.
Ti ventilator | First 10 minutes after birth
  Inspiratory time of a ventilator breath
Ti RIP | First 10 minutes after birth
  Inspiratory time of a spontaneous breath
Ti excess | First 10 minutes after birth
  Calculated: ((Ti ventilator - Ti RIP)/Ti RIP)) x 100
Swing RIP | First 10 minutes after birth
  Amplitude of the RIP curve calculated by subtracting the baseline RIP from the peak RIP curve, which is a surrogate parameter for the patient's respiratory effort.
Number of tactile stimulations and other interventions on the patient | First 10 minutes after birth
  Number of tactile stimulations and other interventions on the patient (e.g. placement of intravenous line, non-invasive administration of surfactant, intubation, chest compression) are documented by video analysis.
Heart rate | First 10 minutes after birth
Oxygen saturation | First 10 minutes after birth
Fraction of inspired oxygen | First 10 minutes after birth

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Warth PP, Ruegger CM, Gaertner VD, Braun W, Molnar K, Brozek J, Poets CF, Springer L. Synchronised Non-Invasive Intermittent Positive Pressure Ventilation in Very Preterm Infants After Birth: A Feasibility Study. Acta Paediatr. 2025 Dec;114(12):3159-3165. doi: 10.1111/apa.70220. Epub 2025 Jul 16. PMID 40665887